## **Official Study Title:**

# **Human Doctors or AI? Evaluating Patient Satisfaction in Urinary Stone Disease Consultations**

### **Statistical Analysis Plan**

NCT number: NCT ID not yet assigned

**Unique Protocol Id: 20243209** 

**Version Date: August 1, 2025** 

#### **Statistical Analysis Plan:**

#### **Descriptive Statistics:**

- Categorical variables: presented as frequency and percentage
- Continuous variables: presented as mean  $\pm$  SD or median (IQR), depending on distribution

#### **Group Comparisons:**

- Primary outcome (CSQ-8 scores): Kruskal-Wallis test to compare satisfaction across all five groups
  - o If significant, post hoc pairwise comparisons with Dunn-Bonferroni correction
- Consultation duration: Kruskal-Wallis test
- Completion rate: Chi-square or Fisher's exact test
- Exploratory analysis: Spearman correlation between satisfaction and age, education level

#### **Significance Level:**

- All tests will be two-sided
- p < 0.05 considered statistically significant